CLINICAL TRIAL: NCT03387280
Title: Electrocardigram Identifying the Culprit Site in Patients With Acute Inferior Myocardial Infarction
Brief Title: ECG Identifying the Culprit Coronary Artery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuan's General Hospital (Other)
Collaborators: Kaohsiung Veterans General Hospital. (Other); Sin-Lau Hospital (Other)
Responsible Party: Principal Investigator, Shoa-Lin Lin, attending Physician, Yuan's General Hospital
Other Study IDs: 20170821B
Record Dates: First submitted 2017-12-21; First posted 2018-01-02 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Acute Myocardial Infarction, of Inferolateral Wall; Acute Myocardial Infarction, of Inferoposterior Wall
Keywords: acute myocardial infarction; electrocardiogram; coronary angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- proximal RCA stenosis: The stenosis site is before the the right ventricular branch of right coronary artery (RCA) according to the coronary angiograms.
- distal RCA stenosis: The stenosis site is after the the right ventricular branch of right coronary artery (RCA) according to the coronary angiograms.
- left circumflex coronary artery stenosis: The stenosis site is located at the left circumflex coronary artery according to the coronary angiograms.

SUMMARY:
Acute myocardial infarction (AMI) usually occurs suddenly and is associated with considerably high mortality rate. The infarct-related artery in inferior wall AMI is usually located at right coronary artery (RCA), less often at left circumflex coronary artery (LCX). Inferior wall AMI occlusive site before the first right ventricular branch of RCA was more frequently associated with right ventricular infarction, which had higher incidence of bradyarrhythmia, shock, and in-hospital death. Early recognition of the site of infarct-related artery especially combination with right ventricular infarction and respond promptly may result in a significant reduction in in-hospital mortality and morbidity. There were several non-invasive methods to predict the culprit site, which including: radioneuclear imaging study, echocardiography or electrocardiogram. Among these methods, electrocardiogram is one of the most simple and convenient tool. Several algorisms have investigated but these algorisms included using leads III, II, I, aVL, V1, V2, V3, V5 and V6, which can only differentiate RCA and LCX lesions but cannot assure whether the culprit site is located at proximal or distal RCA. Thus, the aim of this study is designing a method which is simple and useful in identifying the culprit sites in inferior wall acute myocardial infarction (AMI).

According to the medical record, patients with inferior wall AMI who have no previous history of MI (or the first AMI attack) will be enrolled. These patients are divided into 3 groups from coronary angiography, depending upon the culprit lesion (1) before (proximal) or (2) after (distal) the right ventricular branch of RCA and (3) LCX. A two-step study strategy will be performed to analyze which electrocardiographic variables are capable of discriminating the culprit site of coronary artery. Using the area under the receiver operating characteristic (ROC) curve analysis, we plan to determine which one of the above variables is the most powerful criterion in discriminating the culprit site of coronary artery. Due to the fact that the case number of the first inferior AMI will be limited, this study will be carried out at 3 hospitals in order to collect more cases with the coming year.

DETAILED DESCRIPTION:
Background

Acute myocardial infarction (AMI) usually occurs suddenly and is associated with considerably high mortality rate. The infarct-related artery in inferior wall AMI is usually located at right coronary artery (RCA), less often at left circumflex coronary artery (LCX). [1,2] Inferior wall AMI occlusive site above the first right ventricular branch of RCA was more frequently associated with right ventricular infarction, which had higher incidence of bradyarrhythmia, shock, and in-hospital death.[3-7] Early recognition of the site of infarct-related artery and respond promptly may result in a significant reduction in in-hospital mortality and morbidity.[8-10] Coronary angiography is considered to be the gold standard for determining the culprit site of infarct-related artery, but it is an invasive examination. Additionally, not all hospitals have the facility in performing the cardiac catheterization. There were several non-invasive methods to predict the culprit site including: radioneuclear imaging study, echocardiography or electrocardiogram. Among these methods, electrocardiogram is one of the most simple and useful tools. Several studies have used ST segment elevation in lead III > ST segment elevation in lead II and ST segment depression in lead I, aVL or both to predict that culprit site was located at RCA; ST segment elevation in lead I, aVL, V5 and V6 and ST segment depression in V1, V2 and V3 to predict that the culprit site was located at LCX. [11-24] These electrocardiogram readings including lead III, II, I, aVL, V1, V2, V3, V5 and V6 , which can only differentiate RCA and LCX lesions. If clinicians are intended to know whether the culprit site is located at proximal or distal RCA, further evaluation of the ST segment elevation in leads V1 and V4R,would be needed [25] which makes the algorithm involving too many leads and not so easy to remember. Thus, the aim of this study is designing a method which is simple and useful in identifying the culprit sites in inferior wall acute myocardial infarction (AMI).

Methods

Study Patients:

From review of the medical records, patients suffered from first inferior wall AMI will be enrolled in this study. The diagnosis of acute inferior AMI includes: 1) chest pain > 30 minutes; 2) ST elevation > 1mm in at least two of the three inferior lead (II, III, AVF); and 3) 2-fold increase in serum creatine kinase levels. At least 2 of the above 3 criteria are necessary to confirm the diagnosis. Right ventricular infarction is diagnosed by the presence of an ST-segment elevation of 0.1 mV in the V3R or V4R lead (recorded in all patients with inferior wall MI) in the electrocardiogram performed within 15 minutes after arrival at emergent department. Exclusion criteria include previous AMI or coronary artery bypass surgery, electrocardiographic evidence of bundle branch block, undetermined culprit site by coronary angiography, or first electrocardiogram obtained more than 12 hours after the onset of symptoms. Patient's demographic variables, important risk factors and clinical outcomes including atrioventricular block, arrhythmia, shock, mortality during the first hospital days are recorded.

All patients received dual anti-platelates with aspirin and clopidegrol, and anti-coagulant (low molecular weight heparin or unfractured heparin) regimen. Most of the patients have received primary percutanuous coronary intervention. The GpIIb/IIIa antagonists is administered in all patients.

Electrocardiogarphy:

Standard 12-lead electrocardiogram is performed within 12 hours after onset of chest pain in all study patients. ST-segment deviation from isoelectric line will be measured with a calliper at the point of 80 ms after the J point. The preceding TP-segment is considered as the isoelectric line. The magnitudes of ST-segment deviation in 12-lead electrocardiogram and V4R are also assessed.

Coronary angiography:

Coronary angiography is performed during the first day of admission. The cineangiography films are reviewed by 2 interventional cardiologists who are blinded to the electrocardiographic findings. The culprit artery is defined as total occlusion (Thrombolysis in Myocardial Infarction, TIMI grade 0) or significant stenosis (> 70% diameter stenosis) of RCA or LCX and of their major branches with intraluminal thrombosis or supply to hypokinetic territory. The occlusion site of infarct-related coronary artery determined by coronary angiography is classified into three groups: proximal RCA: lesion proximal to the first right ventricular branch of the RCA; distal RCA: lesion distal to the first right ventricular branch of the RCA; and LCX groups.

Statistical analysis:

The data of electrocardiographic findings, patient's characteristics and clinical outcomes are presented as mean ± standard deviation for continuous variables and frequency distribution for discrete variables. Chi-square analysis is used to assess the association of patients' characteristics with site of culprit lesion. One way ANOVA with Bonferroni post hoc test are used to assess the relation between site of culprit lesion and electrocardiographic findings. The value of P ≤ 0.05 is considered statistically significant. The cut-off point of electrocardiographic criteria for predicting culprit coronary artery is determined by receiver operating characteristic (ROC) curve. The area under the ROC curve represents the diagnostic validity of each cut-off points will be determined and compared.

ELIGIBILITY:
Inclusion Criteria:

* first attacked acute inferior MI patients

Exclusion Criteria:

* those with 1). previous AMI, 2). coronary artery bypass surgery, 3). electrocardiographic evidence of bundle branch block, 4). undetermined culprit site by coronary angiography, 5) first electrocardiogram obtained more than 12 hours after the onset of symptoms.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From review of the medical records, patients suffered from first inferior wall AMI will be enrolled in this study. The diagnosis of acute inferior AMI includes: 1) chest pain > 30 minutes; 2) ST elevation > 1mm in at least two of the three inferior lead (II, III, AVF); and 3) 2-fold increase in serum creatine kinase levels. At least 2 of the above 3 criteria are necessary to confirm the diagnosis.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
determine which criteria is the best one in predicting the culprit site | about 1-2 months
  using ROC curve analysis in the final comparison

CONTACTS AND LOCATIONS:
Overall Officials: Wan Leung, M.D., Study Director — Department of Medical Education & Research of Yuan's General Hospital
Locations (1):
- Yuan's General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Blanke H, Cohen M, Schlueter GU, Karsch KR, Rentrop KP. Electrocardiographic and coronary arteriographic correlations during acute myocardial infarction. Am J Cardiol. 1984 Aug 1;54(3):249-55. doi: 10.1016/0002-9149(84)90176-0. PMID 6464999
- [Background] Berger PB, Ryan TJ. Inferior myocardial infarction. High-risk subgroups. Circulation. 1990 Feb;81(2):401-11. doi: 10.1161/01.cir.81.2.401. No abstract available. PMID 2404629
- [Background] Braat SH, Brugada P, den Dulk K, van Ommen V, Wellens HJ. Value of lead V4R for recognition of the infarct coronary artery in acute inferior myocardial infarction. Am J Cardiol. 1984 Jun 1;53(11):1538-41. doi: 10.1016/0002-9149(84)90575-7. PMID 6731298
- [Background] Braat SH, de Zwaan C, Brugada P, Coenegracht JM, Wellens HJ. Right ventricular involvement with acute inferior wall myocardial infarction identifies high risk of developing atrioventricular nodal conduction disturbances. Am Heart J. 1984 Jun;107(6):1183-7. doi: 10.1016/0002-8703(84)90275-8. PMID 6326559
- [Background] Bueno H, Lopez-Palop R, Bermejo J, Lopez-Sendon JL, Delcan JL. In-hospital outcome of elderly patients with acute inferior myocardial infarction and right ventricular involvement. Circulation. 1997 Jul 15;96(2):436-41. doi: 10.1161/01.cir.96.2.436. PMID 9244209
- [Background] Bueno H, Lopez-Palop R, Perez-David E, Garcia-Garcia J, Lopez-Sendon JL, Delcan JL. Combined effect of age and right ventricular involvement on acute inferior myocardial infarction prognosis. Circulation. 1998 Oct 27;98(17):1714-20. doi: 10.1161/01.cir.98.17.1714. PMID 9788824
- [Background] Mehta SR, Eikelboom JW, Natarajan MK, Diaz R, Yi C, Gibbons RJ, Yusuf S. Impact of right ventricular involvement on mortality and morbidity in patients with inferior myocardial infarction. J Am Coll Cardiol. 2001 Jan;37(1):37-43. doi: 10.1016/s0735-1097(00)01089-5. PMID 11153770
- [Background] Assali AR, Teplitsky I, Ben-Dor I, Solodky A, Brosh D, Battler A, Fuchs S, Kornowski R. Prognostic importance of right ventricular infarction in an acute myocardial infarction cohort referred for contemporary percutaneous reperfusion therapy. Am Heart J. 2007 Feb;153(2):231-7. doi: 10.1016/j.ahj.2006.10.038. PMID 17239681
- [Background] Hamon M, Agostini D, Le Page O, Riddell JW, Hamon M. Prognostic impact of right ventricular involvement in patients with acute myocardial infarction: meta-analysis. Crit Care Med. 2008 Jul;36(7):2023-33. doi: 10.1097/CCM.0b013e31817d213d. PMID 18552681
- [Background] Owens CG, McClelland AJ, Walsh SJ, Smith BA, Stevenson M, Khan MM, Adgey JA. In-hospital percutaneous coronary intervention improves in-hospital survival in patients with acute inferior myocardial infarction particularly with right ventricular involvement. J Invasive Cardiol. 2009 Feb;21(2):40-4. PMID 19182288
- [Background] Assali AR, Herz I, Vaturi M, Adler Y, Solodky A, Birnbaum Y, Sclarovsky S. Electrocardiographic criteria for predicting the culprit artery in inferior wall acute myocardial infarction. Am J Cardiol. 1999 Jul 1;84(1):87-9, A8. doi: 10.1016/s0002-9149(99)00197-6. PMID 10404857
- [Background] Herz I, Assali AR, Adler Y, Solodky A, Sclarovsky S. New electrocardiographic criteria for predicting either the right or left circumflex artery as the culprit coronary artery in inferior wall acute myocardial infarction. Am J Cardiol. 1997 Nov 15;80(10):1343-5. doi: 10.1016/s0002-9149(97)00678-4. PMID 9388111
- [Background] Zimetbaum PJ, Josephson ME. Use of the electrocardiogram in acute myocardial infarction. N Engl J Med. 2003 Mar 6;348(10):933-40. doi: 10.1056/NEJMra022700. No abstract available. PMID 12621138
- [Background] Bayram E, Atalay C. Identification of the culprit artery involved in inferior wall acute myocardial infarction using electrocardiographic criteria. J Int Med Res. 2004 Jan-Feb;32(1):39-44. doi: 10.1177/147323000403200106. PMID 14997704
- [Background] Fiol M, Cygankiewicz I, Carrillo A, Bayes-Genis A, Santoyo O, Gomez A, Bethencourt A, Bayes de Luna A. Value of electrocardiographic algorithm based on "ups and downs" of ST in assessment of a culprit artery in evolving inferior wall acute myocardial infarction. Am J Cardiol. 2004 Sep 15;94(6):709-14. doi: 10.1016/j.amjcard.2004.05.053. PMID 15374771
- [Background] Birnbaum Y, Sclarovsky S, Mager A, Strasberg B, Rechavia E. ST segment depression in a VL: a sensitive marker for acute inferior myocardial infarction. Eur Heart J. 1993 Jan;14(1):4-7. doi: 10.1093/eurheartj/14.1.4. PMID 8432289
- [Background] Kontos MC, Desai PV, Jesse RL, Ornato JP. Usefulness of the admission electrocardiogram for identifying the infarct-related artery in inferior wall acute myocardial infarction. Am J Cardiol. 1997 Jan 15;79(2):182-4. doi: 10.1016/s0002-9149(96)00709-6. PMID 9193020
- [Background] Kabakci G, Yildirir A, Yildiran L, Batur MK, Cagrikul R, Onalan O, Tokgozoglu L, Oto A, Ozmen F, Kes S. The diagnostic value of 12-lead electrocardiogram in predicting infarct-related artery and right ventricular involvement in acute inferior myocardial infarction. Ann Noninvasive Electrocardiol. 2001 Jul;6(3):229-35. doi: 10.1111/j.1542-474x.2001.tb00113.x. PMID 11466142
- [Background] Wong TW, Huang XH, Liu W, Ng K, Ng KS. New electrocardiographic criteria for identifying the culprit artery in inferior wall acute myocardial infarction-usefulness of T-wave amplitude ratio in leads II/III and T-wave polarity in the right V5 lead. Am J Cardiol. 2004 Nov 1;94(9):1168-71. doi: 10.1016/j.amjcard.2004.07.086. PMID 15518613
- [Background] Hasdai D, Birnbaum Y, Herz I, Sclarovsky S, Mazur A, Solodky A. ST segment depression in lateral limb leads in inferior wall acute myocardial infarction. Implications regarding the culprit artery and the site of obstruction. Eur Heart J. 1995 Nov;16(11):1549-53. doi: 10.1093/oxfordjournals.eurheartj.a060776. PMID 8881846
- [Background] Bairey CN, Shah PK, Lew AS, Hulse S. Electrocardiographic differentiation of occlusion of the left circumflex versus the right coronary artery as a cause of inferior acute myocardial infarction. Am J Cardiol. 1987 Sep 1;60(7):456-9. doi: 10.1016/0002-9149(87)90285-2. PMID 3630927
- [Background] Huey BL, Beller GA, Kaiser DL, Gibson RS. A comprehensive analysis of myocardial infarction due to left circumflex artery occlusion: comparison with infarction due to right coronary artery and left anterior descending artery occlusion. J Am Coll Cardiol. 1988 Nov;12(5):1156-66. doi: 10.1016/0735-1097(88)92594-6. PMID 3170958
- [Background] Chia BL, Yip JW, Tan HC, Lim YT. Usefulness of ST elevation II/III ratio and ST deviation in lead I for identifying the culprit artery in inferior wall acute myocardial infarction. Am J Cardiol. 2000 Aug 1;86(3):341-3. doi: 10.1016/s0002-9149(00)00929-2. PMID 10922448
- [Background] Nair R, Glancy DL. ECG discrimination between right and left circumflex coronary arterial occlusion in patients with acute inferior myocardial infarction: value of old criteria and use of lead aVR. Chest. 2002 Jul;122(1):134-9. doi: 10.1378/chest.122.1.134. PMID 12114348
- [Background] Witters PG, Cools FJ. Evaluation of electrocardiographic algorithms in the assessment of the infarct-related artery in acute myocardial infarction. Acta Cardiol. 2006 Aug;61(4):446-53. doi: 10.2143/AC.61.4.2017307. PMID 16970056